CLINICAL TRIAL: NCT01167972
Title: Observational Study on the Management of Patients With Non Small Cell Lung Cancer (NSCLC) Adenocarcinoma Tested for the Activating Mutation of Epidermal Growth Factor Receptor Tyrosine Kinase (EGFR TK)
Brief Title: Observational Study on the Management of Patients With Non Small Cell Lung Cancer Adenocarcinoma
Acronym: MUTACT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OFR-DUM-2010/1
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: M + mutation; Non Small Cell Lung Cancer adenocarcinoma; To determine the proportion of patients with M + mutation status among patients with NSCLC adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The main objective of the study is to determine the proportion of patients with M + mutation status among patients with Non Small Cell Lung Cancer adenocarcinoma.

DETAILED DESCRIPTION:
MSD

ELIGIBILITY:
Inclusion Criteria:

* Patient with lung cancer (Non Small Cell Lung Cancer adenocarcinoma)
* Patient for whom a search for the mutational status of EGFR (EGFR-M +, M- or Mx) has been done or is being analyzed

Exclusion Criteria:

* Assessment of mutational status of EGFR is not done

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with NSCLC adenocarcinoma confirmed by histologyPatient for whom a search for the mutational status of EGFR (EGFR-M +, M- or Mx) has been done or is being analyzed
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The main objective of the study is to determine the proportion of patients with M + mutation status among patients with NSCLC adenocarcinoma | At baseline

SECONDARY OUTCOMES:
Describe the therapeutic management according to the mutational status (EGFR M +, EGFR M- and Mx). | 12 months / At each visit
Describe the therapeutic management of patients with EGFR M +. | 12 months / At each visit
Describe the clinical course of patients EGFR-M +, treated for first-line treatment, and then 2nd line treatment, until 31-AUG-2012 | 12 months / At each visit

CONTACTS AND LOCATIONS:
Overall Officials: Corrine Bernaud, Medical Director, Study Director — AstraZeneca
Locations (101):
- France (101):
  - Research Site, Abbeville
  - Research Site, Aix-en-Provence
  - Research Site, Amilly
  - Research Site, Angers
  - Research Site, Antibes
  - Research Site, Arras
  - Research Site, Aulnay-sous-Bois
  - Research Site, Auxerre
  - Research Site, Bastia
  - Research Site, Bayonne
  - Research Site, Béthune
  - Research Site, Blois
  - Research Site, Bobigny
  - Research Site, Bois-Guillaume
  - Research Site, Bonneville
  - Research Site, Bordeaux
  - Research Site, Boulogne-sur-Mer
  - Research Site, Bourg-en-Bresse
  - Research Site, Brest
  - Research Site, Brive-la-Gaillarde
  - Research Site, Bron
  - Research Site, Caen
  - Research Site, Chalon-sur-Saône
  - Research Site, Chauny
  - Research Site, Clermont-Ferrand
  - Research Site, Colmar
  - Research Site, Compiègne
  - Research Site, Creil
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Douai
  - Research Site, Draguignan
  - Research Site, Fougères
  - Research Site, Gap
  - Research Site, Granville
  - Research Site, La Roche-sur-Yon
  - Research Site, La Rochelle
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Source
  - Research Site, La Tronche
  - Research Site, Le Plessis-Robinson
  - Research Site, Lens
  - Research Site, Levallois-Perret
  - Research Site, Libourne
  - Research Site, Liévin
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Longjumeau
  - Research Site, Lyon
  - Research Site, Mantes-la-Jolie
  - Research Site, Marseille
  - Research Site, Meaux
  - Research Site, Mont-de-Marsan
  - Research Site, Mont-Saint-Martin
  - Research Site, Montauban
  - Research Site, Montivilliers
  - Research Site, Montpellier
  - Research Site, Moulins
  - Research Site, Nevers
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Oloron-Sainte-Marie
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Pessac
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Pontivy
  - Research Site, Pontoise
  - Research Site, Pringy
  - Research Site, Privas
  - Research Site, Redon
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Roanne
  - Research Site, Rouen
  - Research Site, Saint-Aubin-lès-Elbeuf
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Denis
  - Research Site, Saint-Herblain
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Saint-Quentin
  - Research Site, Saintes
  - Research Site, Salouël
  - Research Site, Sarrebourg
  - Research Site, Soissons
  - Research Site, Ste Clotilde
  - Research Site, Ste Feyre
  - Research Site, Strasbourg
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Tours
  - Research Site, Trappes
  - Research Site, Valence
  - Research Site, Vendôme
  - Research Site, Verdun
  - Research Site, Villejuif
  - Research Site, Villenave-d'Ornon
  - Research Site, Yerres